CLINICAL TRIAL: NCT00737581
Title: Posture Responsive Spinal Cord Stimulation Research Study
Brief Title: Spinal Cord Stimulation Research Study
Status: Completed | Type: Observational
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Other Study IDs: 1648
Record Dates: First submitted 2008-08-15; First posted 2008-08-19 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Chronic Low Back and Leg Pain
Keywords: Subject's; response; changes; in spinal; cord; stimulation; during; postural
MeSH Terms: conditions — Cone-Rod Dystrophies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to characterize subjects' response to spinal cord stimulation with postural changes.

ELIGIBILITY:
Inclusion Criteria:

* Be ambulatory
* Be 18 years of age or older
* Have chronic low back pain and/or leg pain due to neuropathic causes
* Be implanted with the Restore or Restore Advanced system for greater than or equal to 3 months
* Be implanted with percutaneous thoracic leads
* Have stable pain control
* Adjust stimulation parameters manually on a regular basis
* Be willing and able to complete protocol requirements
* Be willing and able to provide written informed consent
* Be male or nonpregnant female

Exclusion Criteria:

* Plan to enroll in another clinical study during participation in this study, or currently enrolled in another clinical study
* Be morbidly obese
* Had pain-related surgery in the previous 12 weeks of enrollment or intend to undergo surgery during the period of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients implanted with a spinal cord stimulator.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-08; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Schultz, MD, Principal Investigator — Medical Advanced Pain Specialists; Cristy Schade, MD, Principal Investigator — Center for Pain Control
Locations (2):
- United States (2):
  - Medical Advanced Pain Specialists (MAPS), Edina, Minnesota
  - Center for Pain Control, Garland, Texas